CLINICAL TRIAL: NCT06945926
Title: The Effect of Oxytocin Nasal Spray on Preventing Postoperative Delirium in Elderly Patients Undergoing Orthopedic Surgery：Two-Stage Designs for Phase II Clinical Trials
Brief Title: The Effect of Oxytocin Nasal Spray on Preventing Postoperative Delirium in Elderly Patients Undergoing Orthopedic Surgery
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Diansan Su, Chair of the Department of Anesthesiology, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ZJU2025C045
Record Dates: First submitted 2025-04-08; First posted 2025-04-27 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-03

CONDITIONS: Cervical Spinal Stenosis; Thoracic Spinal Stenosis; Lumbar Spinal Stenosis; Rotator Cuff Injury; Femoral Head Necrosis; Spinal Trauma; Knee Joint Injury
Keywords: Postoperative delirium; elderly orthopedics; oxytocin nasal spray
MeSH Terms: conditions — Spinal Stenosis; Rotator Cuff Injuries; Emergence Delirium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Oxytocin nasal spray given to geriatric orthopedic general anesthesia patients (Experimental): Cases were included according to the inclusion and exclusion criteria, and induction, maintenance and resuscitation were performed according to the standard protocol for general anesthesia.Before the end of anesthesia, the experimenter administered oxytocin nasal spray (Oxytocin) that was 3 sprays in each nostril (4 IU each) for a total of 24 IU. Beginning 1 day postoperatively, administer 24 IU of oxytocin nasal spray 2 times/day in the morning and 24 IU in the evening.Until 7 days after surgery or discharge.
  Interventions: Drug: oxytocin nasal spray

INTERVENTIONS:
Drug: oxytocin nasal spray — Cases were included according to the inclusion and exclusion criteria, and induction, maintenance and resuscitation were performed according to the standard protocol for general anesthesia.Before the end of anesthesia, the experimenter administered oxytocin nasal spray (Oxytocin) that was 3 sprays in each nostril (4 IU each) for a total of 24 IU. Beginning 1 day postoperatively, administer 24 IU of oxytocin nasal spray 2 times/day in the morning and 24 IU in the evening.Until 7 days after surgery or discharge.

SUMMARY:
Postoperative delirium is a delirium that occurs within 7 days after surgery or before hospital discharge. It has been shown that combined POD can increase the incidence of postoperative pulmonary infections, deep vein thrombosis and decubitus ulcers, and increase the incidence of disability and mortality. The incidence of postoperative delirium in geriatric orthopedics is high.

Investigators conduct a prospective clinical study on geriatric orthopedic surgery patients to investigate the effect of oxytocin nasal spray on the prevention of postoperative delirium in geriatric orthopedic surgery. Cases were included according to the inclusion and exclusion criteria, and induction, maintenance and resuscitation were performed according to the standard protocol for general anesthesia. Before the end of surgery, the Investigators administered oxytocin nasal spray (Oxytocin) that was 3 sprays in each nostril (4 IU each) for a total of 24 IU. Beginning 1 day postoperatively, administer 24 IU of oxytocin nasal spray 2 times/day in the morning and in the evening. Until 7 days after surgery or discharge. The sample size are 77 cases in phase I and 143 cases in phase 2, total 220 cases.

ELIGIBILITY:
Elderly patients undergoing orthopedic surgery under general anesthesia

Inclusion criteria:

1. Age ≥ 65 years;
2. Patients who were to undergo elective orthopedic surgery under general anesthesia with tracheal intubation;
3. ASA class I-III;
4. Estimated duration of surgery ≥ 1 hour; (5) The patient himself/herself or his/her legal representative;
5. Informed consent from the patient or legal representative;
6. Proficiency in the use of Chinese language for communication.

Exclusion criteria:

1. Nasal cavity occupation, patients with fillers in the nose
2. Oxytocin allergy;
3. Patients with previous psychiatric and neurological disorders, such as depression, severe central nervous system depression, Parkinson's disease, basal ganglia disease.

   Goldson's disease, basal ganglia lesions, schizophrenia, epilepsy, Alzheimer's disease, myasthenia gravis, and so on;
4. Pregnant and lactating women
5. Patients with severe hepatic insufficiency (Child-Pugh class C);
6. patients with severe renal insufficiency (dialysis is required before surgery)
7. Severe heart failure (METS<4);
8. Preoperative inability to communicate (coma or dementia);
9. Severe preoperative blindness, deafness, or inability to understand Mandarin to complete preoperative delirium screening;
10. Preoperative cognitive impairment as determined by a MoCA evaluation prior to surgery;
11. Patients who are scheduled for 2 surgeries within 7 days of surgery;
12. Patients with bone malignancy
13. Currently participating in other clinical trials.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative delirium within 7 days after surgery. | From the day of surgery to 7 days after surgery.Twice a day after surgery, once in the morning and once in the afternoon
  In the anesthesia recovery room, the CAM-ICU(The Confusion Assessment method for the ICU ) scale was performed 30 min after extubation. Postoperative delirium was measured by the 3D-CAM (The 3-Minute Diagnostic Confusion Assessment Method)scale from postoperative day 1 until postoperative day 7 or before discharge from the hospital. The CAM scale includes four major features: 1. Acute onset or fluctuating changes in condition 2. Inattention 3. Confusion 4. Changes in level of consciousness. Delirium is diagnosed when features 1 and 2 are positive at the same time, and/or features 3 and 4 are positive.

SECONDARY OUTCOMES:
The severity of postoperative delirium | From the day of surgery to 7 days after surgery
  If the patient develops delirium, assess the severity with the MDAS( Memory Disorder Assessment Scale).The total score is 30 points, and the higher the score, the greater the degree of delirium
Length of hospitalization | 1 year
  Recording the duration of hospitalization，Time from admission to discharge

OTHER OUTCOMES:
Time to extubation | Perioperative
  Time from discontinuation of anesthetic drugs to removal of endotracheal tube
Time to PACU stay | Perioperative
  Time from entering the anesthesia recovery room to leaving the anesthesia recovery room
Adverse reactions related to the experimental drugs. | Within 7 days of surgery
  Adverse reactions Occasional symptoms of nasal irritation, nosebleeds, uterine bleeding, uterine hypercontractions and lacrimation
Postoperative complication | Perioperative, up to 1 weeks
  Postoperative complications such as intraoperative knowledge, lung infection, nausea and vomiting
Time of catheter removal and first time out of bed | Perioperative, up to 1 weeks
  Visiting patients daily, inquiring about their condition and keeping timely records

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sawares A, Olver J, Morcos M, Norman T. Oxytocin in old age psychiatry: A systematic review of the safety of using intranasal oxytocin in older adults. Australas Psychiatry. 2025 Feb;33(1):33-44. doi: 10.1177/10398562241291335. Epub 2024 Oct 30. PMID 39474844
- [Background] MacDonald E, Dadds MR, Brennan JL, Williams K, Levy F, Cauchi AJ. A review of safety, side-effects and subjective reactions to intranasal oxytocin in human research. Psychoneuroendocrinology. 2011 Sep;36(8):1114-26. doi: 10.1016/j.psyneuen.2011.02.015. Epub 2011 Mar 23. PMID 21429671
- [Background] Spengler FB, Schultz J, Scheele D, Essel M, Maier W, Heinrichs M, Hurlemann R. Kinetics and Dose Dependency of Intranasal Oxytocin Effects on Amygdala Reactivity. Biol Psychiatry. 2017 Dec 15;82(12):885-894. doi: 10.1016/j.biopsych.2017.04.015. Epub 2017 May 10. PMID 28629540
- [Background] Wang D, Yan X, Li M, Ma Y. Neural substrates underlying the effects of oxytocin: a quantitative meta-analysis of pharmaco-imaging studies. Soc Cogn Affect Neurosci. 2017 Oct 1;12(10):1565-1573. doi: 10.1093/scan/nsx085. PMID 29048602
- [Background] Sarahian N, Khodagholi F, Valian N, Ahmadiani A. Interplay of MeCP2/REST/Synaptophysin-BDNF and intranasal oxytocin influence on Abeta-induced memory and cognitive impairments. Behav Brain Res. 2025 Jan 5;476:115235. doi: 10.1016/j.bbr.2024.115235. Epub 2024 Sep 3. PMID 39236931
- [Background] Jiang J, Zou Y, Xie C, Yang M, Tong Q, Yuan M, Pei X, Deng S, Tian M, Xiao L, Gong Y. Oxytocin alleviates cognitive and memory impairments by decreasing hippocampal microglial activation and synaptic defects via OXTR/ERK/STAT3 pathway in a mouse model of sepsis-associated encephalopathy. Brain Behav Immun. 2023 Nov;114:195-213. doi: 10.1016/j.bbi.2023.08.023. Epub 2023 Aug 28. PMID 37648002
- [Background] Bowen MT. Does peripherally administered oxytocin enter the brain? Compelling new evidence in a long-running debate. Pharmacol Res. 2019 Aug;146:104325. doi: 10.1016/j.phrs.2019.104325. Epub 2019 Jun 21. No abstract available. PMID 31233803
- [Background] Smith AS, Korgan AC, Young WS. Oxytocin delivered nasally or intraperitoneally reaches the brain and plasma of normal and oxytocin knockout mice. Pharmacol Res. 2019 Aug;146:104324. doi: 10.1016/j.phrs.2019.104324. Epub 2019 Jun 22. PMID 31238093
- [Background] Lee MR, Shnitko TA, Blue SW, Kaucher AV, Winchell AJ, Erikson DW, Grant KA, Leggio L. Labeled oxytocin administered via the intranasal route reaches the brain in rhesus macaques. Nat Commun. 2020 Jun 3;11(1):2783. doi: 10.1038/s41467-020-15942-1. PMID 32494001
- [Background] Lee MR, Scheidweiler KB, Diao XX, Akhlaghi F, Cummins A, Huestis MA, Leggio L, Averbeck BB. Oxytocin by intranasal and intravenous routes reaches the cerebrospinal fluid in rhesus macaques: determination using a novel oxytocin assay. Mol Psychiatry. 2018 Jan;23(1):115-122. doi: 10.1038/mp.2017.27. Epub 2017 Mar 14. PMID 28289281
- [Background] Quintana DS, Westlye LT, Alnaes D, Rustan OG, Kaufmann T, Smerud KT, Mahmoud RA, Djupesland PG, Andreassen OA. Low dose intranasal oxytocin delivered with Breath Powered device dampens amygdala response to emotional stimuli: A peripheral effect-controlled within-subjects randomized dose-response fMRI trial. Psychoneuroendocrinology. 2016 Jul;69:180-8. doi: 10.1016/j.psyneuen.2016.04.010. Epub 2016 Apr 22. PMID 27107209
- [Background] Chang SW, Barter JW, Ebitz RB, Watson KK, Platt ML. Inhaled oxytocin amplifies both vicarious reinforcement and self reinforcement in rhesus macaques (Macaca mulatta). Proc Natl Acad Sci U S A. 2012 Jan 17;109(3):959-64. doi: 10.1073/pnas.1114621109. Epub 2012 Jan 3. PMID 22215593
- [Background] Kang YS, Park JH. Brain uptake and the analgesic effect of oxytocin--its usefulness as an analgesic agent. Arch Pharm Res. 2000 Aug;23(4):391-5. doi: 10.1007/BF02975453. PMID 10976589
- [Background] Burkner PC, Williams DR, Simmons TC, Woolley JD. Intranasal Oxytocin May Improve High-Level Social Cognition in Schizophrenia, But Not Social Cognition or Neurocognition in General: A Multilevel Bayesian Meta-analysis. Schizophr Bull. 2017 Oct 21;43(6):1291-1303. doi: 10.1093/schbul/sbx053. PMID 28586471
- [Background] Leppanen J, Ng KW, Tchanturia K, Treasure J. Meta-analysis of the effects of intranasal oxytocin on interpretation and expression of emotions. Neurosci Biobehav Rev. 2017 Jul;78:125-144. doi: 10.1016/j.neubiorev.2017.04.010. Epub 2017 Apr 30. PMID 28467893
- [Background] Shahrestani S, Kemp AH, Guastella AJ. The impact of a single administration of intranasal oxytocin on the recognition of basic emotions in humans: a meta-analysis. Neuropsychopharmacology. 2013 Sep;38(10):1929-36. doi: 10.1038/npp.2013.86. Epub 2013 Apr 10. PMID 23575742
- [Background] Huffmeijer R, van Ijzendoorn MH, Bakermans-Kranenburg MJ. Ageing and oxytocin: a call for extending human oxytocin research to ageing populations--a mini-review. Gerontology. 2013;59(1):32-9. doi: 10.1159/000341333. Epub 2012 Aug 24. PMID 22922544
- [Background] Jesso S, Morlog D, Ross S, Pell MD, Pasternak SH, Mitchell DG, Kertesz A, Finger EC. The effects of oxytocin on social cognition and behaviour in frontotemporal dementia. Brain. 2011 Sep;134(Pt 9):2493-501. doi: 10.1093/brain/awr171. Epub 2011 Aug 22. PMID 21859765
- [Background] Plessow F, Marengi DA, Perry SK, Felicione JM, Franklin R, Holmes TM, Holsen LM, Makris N, Deckersbach T, Lawson EA. Effects of Intranasal Oxytocin on the Blood Oxygenation Level-Dependent Signal in Food Motivation and Cognitive Control Pathways in Overweight and Obese Men. Neuropsychopharmacology. 2018 Feb;43(3):638-645. doi: 10.1038/npp.2017.226. Epub 2017 Sep 20. PMID 28930284
- [Background] Boll S, Almeida de Minas AC, Raftogianni A, Herpertz SC, Grinevich V. Oxytocin and Pain Perception: From Animal Models to Human Research. Neuroscience. 2018 Sep 1;387:149-161. doi: 10.1016/j.neuroscience.2017.09.041. Epub 2017 Sep 28. PMID 28965836
- [Background] van Zuiden M, Frijling JL, Nawijn L, Koch SBJ, Goslings JC, Luitse JS, Biesheuvel TH, Honig A, Veltman DJ, Olff M. Intranasal Oxytocin to Prevent Posttraumatic Stress Disorder Symptoms: A Randomized Controlled Trial in Emergency Department Patients. Biol Psychiatry. 2017 Jun 15;81(12):1030-1040. doi: 10.1016/j.biopsych.2016.11.012. Epub 2016 Dec 8. PMID 28087128
- [Background] Moerkerke M, Daniels N, Tibermont L, Tang T, Evenepoel M, Van der Donck S, Debbaut E, Prinsen J, Chubar V, Claes S, Vanaudenaerde B, Willems L, Steyaert J, Boets B, Alaerts K. Chronic oxytocin administration stimulates the oxytocinergic system in children with autism. Nat Commun. 2024 Jan 2;15(1):58. doi: 10.1038/s41467-023-44334-4. PMID 38167302
- [Background] Sikich L, Kolevzon A, King BH, McDougle CJ, Sanders KB, Kim SJ, Spanos M, Chandrasekhar T, Trelles MDP, Rockhill CM, Palumbo ML, Witters Cundiff A, Montgomery A, Siper P, Minjarez M, Nowinski LA, Marler S, Shuffrey LC, Alderman C, Weissman J, Zappone B, Mullett JE, Crosson H, Hong N, Siecinski SK, Giamberardino SN, Luo S, She L, Bhapkar M, Dean R, Scheer A, Johnson JL, Gregory SG, Veenstra-VanderWeele J. Intranasal Oxytocin in Children and Adolescents with Autism Spectrum Disorder. N Engl J Med. 2021 Oct 14;385(16):1462-1473. doi: 10.1056/NEJMoa2103583. PMID 34644471
- [Background] Striepens N, Kendrick KM, Maier W, Hurlemann R. Prosocial effects of oxytocin and clinical evidence for its therapeutic potential. Front Neuroendocrinol. 2011 Oct;32(4):426-50. doi: 10.1016/j.yfrne.2011.07.001. Epub 2011 Jul 23. PMID 21802441
- [Background] Macdonald K, Macdonald TM. The peptide that binds: a systematic review of oxytocin and its prosocial effects in humans. Harv Rev Psychiatry. 2010 Jan-Feb;18(1):1-21. doi: 10.3109/10673220903523615. PMID 20047458
- [Background] Inouye SK, Westendorp RG, Saczynski JS. Delirium in elderly people. Lancet. 2014 Mar 8;383(9920):911-22. doi: 10.1016/S0140-6736(13)60688-1. Epub 2013 Aug 28. PMID 23992774
- [Background] Scicutella A. The pharmacotherapeutic management of postoperative delirium: an expert update. Expert Opin Pharmacother. 2020 Jun;21(8):905-916. doi: 10.1080/14656566.2020.1738388. Epub 2020 Mar 11. PMID 32156151
- [Background] Alrawashdeh W, Eschweiler J, Migliorini F, El Mansy Y, Tingart M, Rath B. Effectiveness of total knee arthroplasty rehabilitation programmes: A systematic review and meta-analysis. J Rehabil Med. 2021 Jun 2;53(6):jrm00200. doi: 10.2340/16501977-2827. PMID 33846757
- [Background] Aldecoa C, Bettelli G, Bilotta F, Sanders RD, Aceto P, Audisio R, Cherubini A, Cunningham C, Dabrowski W, Forookhi A, Gitti N, Immonen K, Kehlet H, Koch S, Kotfis K, Latronico N, MacLullich AMJ, Mevorach L, Mueller A, Neuner B, Piva S, Radtke F, Blaser AR, Renzi S, Romagnoli S, Schubert M, Slooter AJC, Tommasino C, Vasiljewa L, Weiss B, Yuerek F, Spies CD. Update of the European Society of Anaesthesiology and Intensive Care Medicine evidence-based and consensus-based guideline on postoperative delirium in adult patients. Eur J Anaesthesiol. 2024 Feb 1;41(2):81-108. doi: 10.1097/EJA.0000000000001876. Epub 2023 Aug 30. PMID 37599617
- [Background] Qureshi O, Arthur ME. Recent advances in predicting, preventing, and managing postoperative delirium. Fac Rev. 2023 Jul 28;12:19. doi: 10.12703/r/12-19. eCollection 2023. PMID 37529149
- [Background] Li T, Li J, Yuan L, Wu J, Jiang C, Daniels J, Mehta RL, Wang M, Yeung J, Jackson T, Melody T, Jin S, Yao Y, Wu J, Chen J, Smith FG, Lian Q; RAGA Study Investigators. Effect of Regional vs General Anesthesia on Incidence of Postoperative Delirium in Older Patients Undergoing Hip Fracture Surgery: The RAGA Randomized Trial. JAMA. 2022 Jan 4;327(1):50-58. doi: 10.1001/jama.2021.22647. PMID 34928310
- [Background] Heymann A, Radtke F, Schiemann A, Lutz A, MacGuill M, Wernecke KD, Spies C. Delayed treatment of delirium increases mortality rate in intensive care unit patients. J Int Med Res. 2010 Sep-Oct;38(5):1584-95. doi: 10.1177/147323001003800503. PMID 21309472
- [Background] Milisen K, Van Grootven B, Hermans W, Mouton K, Al Tmimi L, Rex S, Detroyer E. Is preoperative anxiety associated with postoperative delirium in older persons undergoing cardiac surgery? Secondary data analysis of a randomized controlled trial. BMC Geriatr. 2020 Nov 18;20(1):478. doi: 10.1186/s12877-020-01872-6. PMID 33208091
- [Background] Witlox J, Eurelings LS, de Jonghe JF, Kalisvaart KJ, Eikelenboom P, van Gool WA. Delirium in elderly patients and the risk of postdischarge mortality, institutionalization, and dementia: a meta-analysis. JAMA. 2010 Jul 28;304(4):443-51. doi: 10.1001/jama.2010.1013. PMID 20664045
- [Background] Park SK, Lim T, Cho H, Yoon HK, Lee HJ, Lee JH, Yoo S, Kim JT, Kim WH. Comparative effectiveness of pharmacological interventions to prevent postoperative delirium: a network meta-analysis. Sci Rep. 2021 Jun 7;11(1):11922. doi: 10.1038/s41598-021-91314-z. PMID 34099790
- [Background] Meagher D. Motor subtypes of delirium: past, present and future. Int Rev Psychiatry. 2009 Feb;21(1):59-73. doi: 10.1080/09540260802675460. PMID 19219713
- [Background] Olin K, Eriksdotter-Jonhagen M, Jansson A, Herrington MK, Kristiansson M, Permert J. Postoperative delirium in elderly patients after major abdominal surgery. Br J Surg. 2005 Dec;92(12):1559-64. doi: 10.1002/bjs.5053. PMID 16231283